CLINICAL TRIAL: NCT01603576
Title: Safety and Feasibility Study of a Prototype Suprachoroidal Retinal Prosthesis for Vision Restoration
Brief Title: Pilot Study of a Suprachoroidal Retinal Prosthesis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Center for Eye Research Australia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BVA_0001; 090/2012 (Registry Identifier: Therapeutics Goods Administration, Australia)
Record Dates: First submitted 2012-05-18; First posted 2012-05-22 (Estimated); Last update posted 2016-11-16 (Estimated); Status verified 2016-11

CONDITIONS: Retinitis Pigmentosa; Choroideremia
MeSH Terms: conditions — Retinitis Pigmentosa; Choroideremia

ARMS (1):
- Suprachoroidal retinal prosthesis (Experimental)
  Interventions: Device: Prototype wide view suprachoroidal retinal prosthesis

INTERVENTIONS:
Device: Prototype wide view suprachoroidal retinal prosthesis — Manufacturer = Bionics Institute, Australia

SUMMARY:
This study will be an initial proof of concept study, to evaluate safety and efficacy of a prototype suprachoroidal retinal implant

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older
* Either gender
* A confirmed history of outer retinal degenerative disease such as retinitis pigmentosa or choroideremia
* Remaining visual acuity of bare light perception or less in both eyes
* Functional inner retina (ganglion cells and optic nerve), as shown by the ability to perceive light and/or a measurable corneal electrically evoked visual response
* A history of at least 10 years of useful form vision in the worse seeing eye
* Must be willing and able to comply with the testing and follow-up protocol demands (preferably residing within 1.5 hours of the investigational site)

Exclusion Criteria:

* Optic nerve disease (history of glaucoma of more than 1 month, or history of any other optic neuropathy)
* Diseases of the inner retina including, but not limited to, central retinal artery or vein occlusion (CRAO, CRVO), end stage diabetic retinopathy, retinal detachment, traumatic retinal damage, infectious retinal disease, inflammatory retinal disease.
* Inability to visualise the retina due to corneal or other ocular media opacities (corneal degenerations, dense cataracts, trauma, lid malpositions)
* Any ocular condition that predisposes the subject to rubbing their eyes
* Cognitive deficiencies, including dementia or progressive neurological disease
* Psychiatric disorders, including depression, as diagnosed by a qualified psychologist
* Deafness or significant hearing loss
* Inability to speak or understand English
* Pregnancy
* Presence of a cochlear implant
* Subject enrolled in another investigational drug or device trial for the treatment of their ocular condition
* Poor general health, which would exclude them from obtaining a general anaesthetic
* Unrealistic expectations of the bionic eye device

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2012-05; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Safety | 18 months
  Number of device-related serious adverse events

SECONDARY OUTCOMES:
Ability to perceive visual percepts during device stimulation | 18 months
  Number of participants able to perceive phosphenes when the device is stimulated

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Burkitt, PhD, Study Director — Bionic Vision Australia; Robyn Guymer, MBBS, PhD, Principal Investigator — Center for Eye Research Australia
Locations (2):
- Australia (2):
  - Nicta / Data61, Canberra, Australian Capital Territory
  - Centre for Eye Research Australia, East Melbourne, Victoria

REFERENCES:
- [Derived] Shivdasani MN, Sinclair NC, Gillespie LN, Petoe MA, Titchener SA, Fallon JB, Perera T, Pardinas-Diaz D, Barnes NM, Blamey PJ; Bionic Vision Australia Consortium. Identification of Characters and Localization of Images Using Direct Multiple-Electrode Stimulation With a Suprachoroidal Retinal Prosthesis. Invest Ophthalmol Vis Sci. 2017 Aug 1;58(10):3962-3974. doi: 10.1167/iovs.16-21311. PMID 28793152
- [Derived] Petoe MA, McCarthy CD, Shivdasani MN, Sinclair NC, Scott AF, Ayton LN, Barnes NM, Guymer RH, Allen PJ, Blamey PJ; Bionic Vision Australia Consortium. Determining the Contribution of Retinotopic Discrimination to Localization Performance With a Suprachoroidal Retinal Prosthesis. Invest Ophthalmol Vis Sci. 2017 Jun 1;58(7):3231-3239. doi: 10.1167/iovs.16-21041. PMID 28660276
- [Derived] Slater KD, Sinclair NC, Nelson TS, Blamey PJ, McDermott HJ; Bionic Vision Australia Consortium. neuroBi: A Highly Configurable Neurostimulator for a Retinal Prosthesis and Other Applications. IEEE J Transl Eng Health Med. 2015 Jul 13;3:3800111. doi: 10.1109/JTEHM.2015.2455507. eCollection 2015. PMID 27170910
- [Derived] Ayton LN, Blamey PJ, Guymer RH, Luu CD, Nayagam DA, Sinclair NC, Shivdasani MN, Yeoh J, McCombe MF, Briggs RJ, Opie NL, Villalobos J, Dimitrov PN, Varsamidis M, Petoe MA, McCarthy CD, Walker JG, Barnes N, Burkitt AN, Williams CE, Shepherd RK, Allen PJ; Bionic Vision Australia Research Consortium. First-in-human trial of a novel suprachoroidal retinal prosthesis. PLoS One. 2014 Dec 18;9(12):e115239. doi: 10.1371/journal.pone.0115239. eCollection 2014. PMID 25521292
- [Derived] Shivdasani MN, Sinclair NC, Dimitrov PN, Varsamidis M, Ayton LN, Luu CD, Perera T, McDermott HJ, Blamey PJ; Bionic Vision Australia Consortium. Factors affecting perceptual thresholds in a suprachoroidal retinal prosthesis. Invest Ophthalmol Vis Sci. 2014 Sep 9;55(10):6467-81. doi: 10.1167/iovs.14-14396. PMID 25205858